CLINICAL TRIAL: NCT04078009
Title: Nasal Allergen Challenge: Standardisation as a Surrogate for Hay Fever
Brief Title: Standardising Nasal Allergen Challenge in Adult With Hay Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 19IC5338
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Allergic Rhinitis
Keywords: Grass pollen allergy; Hayfever; Atopy; Allergic rhinitis; Nasal allergen challenge
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: This is a single group study assessing symptoms scores 4 weeks between the two assessments (Grazax NAC and Aquagen NAC) performed to avoid any carry-over effects of this cross-over design.
Masking Description: An open labelled randomised to either start with Aquagen or Grazax NAC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquagen (Starts with Aquagen and finish with Grazax) (Experimental): In order to explore a possible order effect with the challenges, in this single group cross-over trial, participants will be randomised (by computer-generated randomisation) to receive either Aquagen or Grazax as the first challenge, followed by the other allergen extract at the second challenge a minimum of 4 weeks later.
  Interventions: Diagnostic Test: Aquagen
- Grazax (Starts with Grazax and finish with Aquagen) (Experimental): In order to explore a possible order effect with the challenges, in this single group cross-over trial, participants will be randomised (by computer-generated randomisation) to receive either Aquagen or Grazax as the first challenge, followed by the other allergen extract at the second challenge a minimum of 4 weeks later.
  Interventions: Diagnostic Test: Grazax

INTERVENTIONS:
Diagnostic Test: Aquagen — To compare the clinical allergic response after direct installation of an aqueous solution of Aquagen Timothy Grass pollen extract via nasal allergen challenge with the clinical allergic response after direct installation of an aqueous solution of Grazax Timothy Grass lyophilisate tablets via nasal allergen challenge in grass pollen allergic individuals.
  Other Names: Grazax Timothy Grass lyophilisate tablet
  Arms: Aquagen (Starts with Aquagen and finish with Grazax)
Diagnostic Test: Grazax — To compare the clinical allergic response after direct installation of an aqueous solution of Aquagen Timothy Grass pollen extract via nasal allergen challenge with the clinical allergic response after direct installation of an aqueous solution of Grazax Timothy Grass lyophilisate tablets via nasal allergen challenge in grass pollen allergic individuals.
  Arms: Grazax (Starts with Grazax and finish with Aquagen)

SUMMARY:
Hay fever affects 1 in 4 of the UK population and has significant effects on the quality of life of sufferers. Allergy to grass pollen is the most common cause. A detailed understanding of the mechanisms involved during allergic reactions to pollens in hay fever sufferers may provide improvements in diagnosis, drug treatment and assessment of their response to treatment.

Controlled exposures to allergens such as grass pollen can provide important information on the mechanisms of allergic inflammation and may be used to assess the success of anti-allergy treatments.

Nasal allergen challenge (NAC) is a useful tool in the investigation of allergic rhinitis, including grass pollen-induced seasonal allergic rhinitis (hay fever). NAC is performed by installation of a very small amount of grass pollen extract into the nose in order to reproduce mild and short-lived symptoms such as nasal itch, sneezing, runny nose and nasal congestion that you experience in a more severe form during natural exposure to grass pollen during the summer. Nasal allergen challenge has allowed us to explore the mechanism of hay fever and to provide a rapid and reliable method for investigating new potential treatments for hay fever.

Nasal allergen Challenge is a very well-standardised and safe procedure that has been performed within the department of Allergy and Clinical Immunology at Imperial College and Royal Brompton Hospital for many years.

Unfortunately the grass pollen extract ('Aquagen') that we have routinely used for nasal challenge has been discontinued and is therefore no longer available. The present study involves testing an alternative source of the grass pollen extract in the form of 'Grazax' which is a freeze-dried tablet that is highly standardised and should enable us to give an identical amount of grass pollen extract for the purpose of nasal challenge. We plan a 'head-to-head' comparison of the two extracts in nasal challenge in order to confirm that the two sources of allergen are equivalent thereby enabling us to use Grazax as the source of grass pollen extract for our nasal challenge studies in the future.

DETAILED DESCRIPTION:
Nasal allergen challenge (NAC) is a useful tool in the investigation of allergic rhinitis, including grass pollen-induced seasonal allergic rhinitis (hay fever). We have experience in using NAC to investigate the clinical and immunological effects of allergen exposure and in using NAC as a surrogate outcome to assess the efficacy of treatments for allergic rhinitis. The procedure is safe and well tolerated. In order for NAC to be a valid tool, it is essential that the allergen extracts used are standardised in terms of concentration and stability in solution. We have previously used an extract of Timothy Grass (Phleum pratense) pollen, Aquagen (ALK-Abello, Denmark). Aquagen is supplied as a dry powder, to be reconstituted prior to use by dissolving in an albumin-based diluent. Unfortunately, Aquagen production has been discontinued, but the identical allergen is now available as Timothy Grass lyophilisate tablet, Grazax (ALK-Abello), an approved and licensed product for treatment of severe seasonal allergic rhinitis. Grazax consists of purified, freeze-dried Timothy Grass pollen extract, plus only three excipients, gelatin (from fish), mannitol and sodium hydroxide. Preliminary investigations have shown that Grazax tablets can be dissolved in saline to produce identical concentrations of allergen to Aquagen, with the same stability profile in vitro. We anticipate therefore, that the clinical effect when used for nasal allergen challenges would be equivalent to the use of Aquagen for a given allergen concentration. In this study we intend to confirm that nasal symptoms produced during the NAC with either Aquagen or Grazax will be equivalent. We will recruit volunteers with grass pollen-induced hay fever to undergo NAC with each allergen source, sequentially. In an open, randomised-order, cross-over study. The primary outcome will be patient-reported nasal symptoms (according to a standardised scoring system) in the 60 minutes after each nasal challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 65 years.
2. A clinical history of moderate-severe grass pollen-induced allergic rhino conjunctivitis for at least 2 years with peak symptoms from mid-May to mid-July.
3. Positive skin prick test response, defined as wheal diameter ≥ 5 mm, to timothy grass pollen.
4. For women of childbearing age, a negative urine pregnancy test at the time of screening and willingness to use an effective form of contraception for the duration of involvement in the study.
5. The ability to give informed consent and comply with study procedures.

Exclusion Criteria:

1. History of previous grass pollen allergen immunotherapy at any time in the past.
2. Pre-bronchodilator FEV1 < 70% of predicted value at screening.
3. A clinical history of symptomatic allergic rhinitis and/or asthma caused by an allergen other than grass pollen to which the participant is regularly exposed either seasonally (eg. tree pollen, weed pollen and moulds) or perennially (house dust mite, cat, dog dander).
4. Perennial asthma requiring regular inhaled corticosteroids.
5. History of emergency visit or hospital admission for asthma in the previous 12 months.
6. History of chronic obstructive pulmonary disease
7. History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment.
8. History of chronic sinusitis, defined as sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, ear pain, pressure, or fullness.
9. At screening visit, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
10. History of life-threatening anaphylaxis or angioedema.
11. Ongoing systemic immunosuppressive treatment.
12. The use of any investigational drug within 30 days of the screening visit.
13. The presence of any medical condition that the investigator deems incompatible with participation in the study.
14. History of fish allergy with positive skin test and/or positive specific IgE test to vertebrate/finned fish (due to potential fish allergen exposure from fish-gelatin in Grazax).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Total nasal symptoms scores after nasal allergen challenge | 60 minutes
  To compare the total nasal symptom score at one hour after grass pollen nasal allergen challenge in Aquagen group versus Grazax group. Score ranges from 0-12 points. Higher score is more severe symptoms.

SECONDARY OUTCOMES:
Peak nasal inspiratory flow | Baseline, 60 minutes
  Area under the curve for peak nasal inspiratory flow (PNIF) (delta PNIF change from baseline) 0-60 minutes post NAC. Bland Altman plots will also be utilized for the analysis of the secondary endpoint of delta PNIF AUC.
Incidence of Adverse Events | 48 hours
  To evaluate the safety and tolerability of the nasal allergen challenge administered with each allergen source (Aquagen or Grazax). Participant and investigator reported adverse events potentially related to study procedures, including nasal allergen challenge, will be recorded (typical symptoms of hay fever following nasal allergen challenge lasting less than 24 hours will not be considered adverse events). Frequency of adverse events will be tabulated by event, system organ class, severity, and procedure relatedness as per CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Stephen Durham, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No